CLINICAL TRIAL: NCT06429033
Title: A Phase 1 Controlled Study to Evaluate the Safety and Tolerability of Intradermal Administered Purified Exosome Product (PEP) in Healthy Adults
Brief Title: Purified Exosome Product (PEP) Injected Into the Hypodermis
Acronym: PEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinical Testing of Beverly Hills (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PEP-23-002
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): A single dose of PEP (Purified Exosome Product) in Lactated Ringers at doses of 1 vial (75 mg) (Low Dose/Cohort 1) or 2 vials (150 mg) (Target Dose/Cohort 2) will be injected intradermally into the hypodermis of a 5 cm by 10 cm section of abdomen (to the right of the umbilicus) that is planned for removal during abdominoplasty surgery. The solution will be injected into the hypodermis in retrograde linear threads.
  Interventions: Drug: PEP (Purified Exosome Product)

INTERVENTIONS:
Drug: PEP (Purified Exosome Product) — Injection of PEP into hypodermis of abdomen

SUMMARY:
This clinical trial aims to characterize the safety, tolerability, and histological profile of PEP (Purified Exosome Product) when injected into the hypodermis of healthy adults. The main questions this study aims to answer are:

Is PEP safe and tolerable when injected into the hypodermis of healthy adults?

Subjects will serve as their own control and researchers will compare PEP to Control to see if PEP is safe.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, within-subject, controlled, single center, open-label study. Up to 9 healthy adult participants with planned elective body reduction surgery to remove excess skin on the abdomen in 30-45 days will be enrolled and injected with a single dose of PEP Drug Product reconstituted in Lactated Ringers (USP) solution in a defined area of the abdominal hypodermis. Similar tissue from the participant's contralateral side of the abdomen will serve as the control. Excised tissue will be harvested and analyzed for key biological markers for skin quality and senescence such as collagen and elastin. The primary goal of this investigator-initiated study is to determine safety of subcutaneous PEP Drug Product when reconstituted in Lactated Ringers solution. Safety data will be collected with frequent monitoring for adverse events, laboratory testing, vital signs, and ECGs.

Note: The decision to undergo abdominoplasty will be made outside of this study and data/safety in the plastic surgery procedure for abdominoplasty, other than informed consent, will not be a collected as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants aged 18-65 (inclusive)
* Capacity to sign informed consent.
* Planned elective body reduction surgery to remove excess skin on the abdomen in ≥ 12 to ≤ 18 weeks
* Participant is judged, by the clinical investigator, to be healthy as evidenced by lack of clinically significant abnormal findings on medical history, physical examination, vital signs, and clinical laboratory tests.
* Participant should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods (laser devices, topical prescriptions, or other known hair growth treatments) in the treatment area during the entire study period.
* Females of childbearing potential must be using an approved method of birth control for the past month and during the entire study period. Participants who can become pregnant will undergo a pregnancy test prior to treatment.

Exclusion Criteria:

* Participants with clinically abnormal hematology, serum chemistries, or screening laboratory results as reviewed by the clinical investigator.
* Known history of MRSA (methicillin-resistant staphylococcus aureus).
* Known history of COVID-19 infection in past 6 months.
* COVID vaccine or booster dose within past 12 weeks.
* Participants who are positive for hepatitis B surface antigen (HbsAg), hepatitis C antibody, or HIV.
* History of antibiotic use in past 12 weeks.
* Major surgery in past 3 months.
* If taking hormone replacement therapy or hormones for birth control, dose must be stable for at least 6 months prior to study entry.
* Current or regular use of corticosteroids during the previous 4 weeks, excluding inhaled or topical steroids outside of the planned treatment area.
* Known sensitivity/allergy to study product ingredients.
* Pregnancy and nursing or lactating.
* Sexually active women of childbearing potential who are unwilling to use approved contraception method for three months after receiving dose of investigational drug.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, history of any malignancies or metabolic disease that is, in the opinion of the investigator, not stabilized or may otherwise impact the results of the study.
* Participants with hepatic impairment
* Participants with poorly controlled diabetes mellitus (HbA1C ≥ 8%).
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Any surgery or treatment such as laser or chemicals in the treatment area within 6 months prior to treatment
* History of excessive UV exposure (e.g., frequent sunburn, use of tanning beds, or prolonged outdoor activities without adequate sun protection)
* Any medical condition that in the opinion of the investigator, such condition would compromise the safety of the participant or quality of the study data.
* Current, or past participation in a clinical trial within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Safety: Dose limiting toxicities | 14-days
  The number of subjects with acute dose-limiting toxicities
Maximum Tolerated Dose | 14-days
  The maximum tolerated dose determined by testing increasing doses of PEP
Incidence of withdrawls from the study due to treatment-emergent adverse events | 30 days
  The number of subjects withdrawn from the study due to treatment-emergent adverse events
Incidence of Treatment-Emergent Adverse Events | 30 days
  The number of subjects experiencing treatment emergent adverse events
Common Treatment Responses | 14-days
  The number of subjects experiencing injection site reactions as noted in the patient diary
Laboratory Changes | 30 days
  The number of subjects with changes and shifts from baseline in laboratory measurements
Application Site Reactions | 14 days
  The number of subjects experiencing changes from baseline in treatment application site reactions

CONTACTS AND LOCATIONS:
Overall Officials: John H Joseph, MD, Principal Investigator — Clinical Testing Center
Locations (1):
- Clinical Testing of Beverly Hills, Encino, California, United States

IPD SHARING:
Plan to Share IPD: No